CLINICAL TRIAL: NCT04007523
Title: Recommendations and Alerting for Delirium Alleviation in Real-Time (RADAR): a Pilot Randomized Controlled Trial
Brief Title: Recommendations and Alerting for Delirium Alleviation in Real-Time (RADAR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The Claude D. Pepper Older Americans Independence Centers (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Phillip Vlisides, Assistant Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00165251; 5P30AG024824-15 (NIH)
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Delirium
Keywords: Caregivers; Clinical Decision Support Systems; Cognitive Dysfunction; Confusion; Delirium; Feasibility Studies; Geriatric Assessment; Neurocognitive Disorders
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Confusion; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care Group (No Intervention): Usual care per surgical ward standards
- HELP Support System (Experimental): This arm will receive the HELP Support System intervention only
  Interventions: Behavioral: HELP Support System
- Family Support System (Experimental): This arm will receive the Family Support system intervention only
  Interventions: Behavioral: Family Support System
- Combined Support Systems (Experimental): Participants randomized to this arm will receive both HELP- and family-based support system interventions
  Interventions: Behavioral: Family Support System; Behavioral: HELP Support System

INTERVENTIONS:
Behavioral: Family Support System — Family members and/or caregivers of patients will receive pagers, and alerts will provide recommendations for daily delirium screening and therapeutic activities. Protocols with associated activities will be provided to family members.
  Arms: Combined Support Systems; Family Support System
Behavioral: HELP Support System — A postoperative page will be sent, on behalf of participants, to the on-call HELP staff. The page will request early evaluation and enhanced therapeutic protocols for delirium prevention.
  Arms: Combined Support Systems; HELP Support System

SUMMARY:
This is a pilot randomized controlled trial that will test whether a multicomponent decision support system will improve the postoperative environment for neurocognitive and clinical recovery in older, high-risk surgical patients. Decision support systems will be tested that provide targeted alerts and recommendations to the Hospital Elder Life Program and family members for delirium prevention.

DETAILED DESCRIPTION:
Delirium is a distressing and common surgical complication, affecting approximately 20-50% of older surgical patients. Postoperative delirium is associated with increased mortality, cognitive and functional decline, and healthcare resource utilization. Prevention programs have been tested with variable success, but the Hospital Elder Life Program (HELP) has consistently been demonstrated to reduce the incidence and impact of delirium. However, substantial resources are needed for program operations, and complementary support systems may help with patient triage and assessment. Family members and caretakers may be able to provide supplementary support with delirium screening and prevention via targeted, therapeutic activities. Thus, an automated postoperative paging system, which elicits additional, focused support from HELP and family members, may augment delirium prevention activities and reduce associated risk.

The primary objectives of this study are to determine whether pager-based clinical decision support systems bolster HELP- and family-based therapeutic activities. A secondary objective will be to identify facilitators and barriers to delivering therapeutic interventions for both HELP and family members. Overall, this pilot trial will test the hypothesis that a multicomponent decision support system will improve the postoperative environment for neurocognitive and clinical recovery in older, high-risk surgical patients. Patients (n=60) will be randomized to one of four groups in a factorial design: usual care (n=15), HELP-based paging system (n=15), family-based paging system (n=15), or both HELP- and family-based paging system (n=15). The support systems will consist of automated pager alerts to the HELP program and/or family members and caretakers, depending on group allocation, for providing additional delirium evaluation and therapeutic prevention activities. Outcomes will include various clinical, neurocognitive, and functional measures, and performance metrics will be collected regarding HELP- and family-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years of age
* Major non-cardiac, non-intracranial neurologic, and non-major vascular surgery
* Anticipated length of stay at least 72 hours
* At least one family member, or caretaker, available on each of the first three postoperative days for trial operations

Exclusion Criteria:

* Emergency surgery
* Severe cognitive impairment (precluding ability to perform delirium assessments)
* Planned postoperative ICU admission
* Non-English speaking

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip E Vlisides, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical School, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vlisides PE, Runstadler N, Martinez S, Ragheb JW, Mentz G, Leis A, Schoettinger A, Hickey K, McKinney A, Brooks J, Zierau M, Norcott A, Mody L, Inouye SK, Avidan MS, Min L. Feasibility of Alerting Systems and Family Care Partner Support for Postoperative Delirium Prevention. J Neurosurg Anesthesiol. 2025 Oct 1;37(4):361-370. doi: 10.1097/ANA.0000000000001016. Epub 2024 Dec 19. PMID 39696755
- [Derived] Vlisides PE, Ragheb JW, Leis A, Schoettinger A, Hickey K, McKinney A, Brooks J, Zierau M, Norcott A, Yang S, Avidan MS, Min L. Recommendations and Alerting for Delirium Alleviation in Real-Time (RADAR): Protocol for a pilot randomized controlled trial. F1000Res. 2019 Sep 24;8:1683. doi: 10.12688/f1000research.20597.2. eCollection 2019. PMID 32934794

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Withdrawn (n=3); surgery cancelled (n=2), staff availability (n=1)
Period: Overall Study
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Started (Of note: the Withdrawals by Subjects in this section occurred after trial arm allocation and were separate from the n=3 withdrawals listed above in the Pre-assignment Details.) | 15 | 12 | 14 | 16
Completed | 15 | 10 | 11 | 13
Not Completed | 0 | 2 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — ICU Transfer | 0 | 1 | 0 | 0
Not completed — COVID hospital closure | 0 | 0 | 1 | 2
Not completed — Surgery cancelled | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems | Total
Number analyzed (Participants) | 15 | 10 | 11 | 13 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (4) | 76 (5) | 78 (4) | 77 (7) | 77 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 6 | 7 | 26
  Male | 6 | 6 | 5 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 10 | 10 | 13 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 15 | 9 | 10 | 13 | 47
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Delirium
Description: Any positive delirium screen (yes/no) as determined by the long-form Confusion Assessment Method (n, 0-19)
Time Frame: morning postoperative day one through afternoon of postoperative day three
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 15 | 10 | 11 | 13
Participants | 3 | 3 | 1 | 2
Statistical Analysis 1: Comparison: Usual Care Group vs HELP Support System; Test type: Other — Fisher's Exact Test; p = 0.653, Fisher Exact
Statistical Analysis 2: Comparison: Usual Care Group vs Family Support System; Test type: Other — Fisher's Exact Test; p = 0.614, Fisher Exact
Statistical Analysis 3: Comparison: Usual Care Group vs Combined Support Systems; Test type: Other — Fisher's Exact Test; p = 0.999, Fisher Exact

2. Secondary Outcome: Delirium Severity
Description: For any patient with a completed delirium assessment, the associated severity score will be recorded using the Confusion Assessment Method Long Form Severity Score (n, 0-19, with higher number indicating more severe delirium)
Time Frame: morning postoperative day one through afternoon of postoperative day three
Population: Delirium severity data are derived from all available, completed delirium assessments within each group.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 15 | 10 | 11 | 13
score on a scale | 2 [0 to 3] | 1 [0 to 3] | 3 [1 to 5] | 2 [1 to 2]

3. Secondary Outcome: Depressive Symptoms as Assessed by Hospitalized Anxiety and Depression Scale (HADS-D)
Description: Incidence (%) of positive screens (score ≥8) using the Hospitalized Anxiety and Depression Scale (HADS-D) (n, 0-21, 0 = normal, 21 = presence of severe depression symptoms)
Time Frame: baseline through postoperative day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 12 | 8 | 7 | 11
Participants | 1 | 1 | 1 | 1

4. Secondary Outcome: Anxiety Symptoms as Assessed by Hospitalized Anxiety and Depression Scale (HADS-A)
Description: Incidence (%) of positive screens (score ≥8) using the Hospitalized Anxiety and Depression Scale (HADS-A) (n, 0-21, 0 = normal, 21 = presence of severe anxiety symptoms)
Time Frame: baseline through postoperative day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 13 | 8 | 7 | 11
Participants | 2 | 1 | 0 | 0

5. Secondary Outcome: Falls
Description: Proportion of patients in each group (%) experiencing at least one fall
Time Frame: morning postoperative day one through afternoon of postoperative day three
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 15 | 10 | 11 | 13
Participants | 0 | 1 | 0 | 0

6. Secondary Outcome: Length of Hospital Stay
Description: Total number of days (n) spent in the hospital, up to 30 days
Time Frame: morning of surgery until day of hospital discharge, up to 30 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 15 | 10 | 11 | 13
Days | 4 [2 to 5] | 5 [3 to 6] | 4 [3 to 7] | 4 [3 to 7]

7. Secondary Outcome: Discharge Disposition
Description: Proportion of patients in each group (%) discharged somewhere other than home (e.g., Long-Term Care Facility), up to 30 days
Time Frame: day of hospital discharge, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 15 | 10 | 11 | 13
Participants | 2 | 1 | 3 | 1

8. Secondary Outcome: Delayed Discharge - Cognitive Impairment
Description: Proportion of patients in each group (%) experiencing delayed discharge, with the documented reason as cognitive impairment
Time Frame: day of hospital discharge, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 15 | 10 | 11 | 13
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: New Non-surgical Site Infection
Description: Incidence (%) of any new non-surgical site infection while hospitalized
Time Frame: morning of surgery until day of hospital discharge, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 15 | 10 | 11 | 13
Participants | 0 | 1 | 1 | 2

10. Secondary Outcome: Multidrug Resistant Organism Colonization
Description: Incidence (%) of any new multidrug resistant organism colonization
Time Frame: morning postoperative day one through 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 15 | 10 | 11 | 13
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Mortality
Description: Incidence (%)
Time Frame: within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
Number analyzed (Participants) | 15 | 10 | 11 | 13
Participants | 1 | 0 | 0 | 0

12. Other Pre Specified Outcome: HELP - Duration of Time
Description: Cumulative length of time spent with HELP team members
Time Frame: postoperative day one through postoperative day three
Reporting Status: Not Posted

13. Other Pre Specified Outcome: HELP - Visitation
Description: Proportion of patients successfully visited by the program
Time Frame: postoperative day one through postoperative day three
Reporting Status: Not Posted

14. Other Pre Specified Outcome: HELP - Time to Evaluation
Description: Time until initial HELP evaluation
Time Frame: postoperative day one through postoperative day three
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Family Intervention - Duration of Time
Description: Cumulative duration of time spent with family members/caretakers at the bedside
Time Frame: postoperative day one through postoperative day three
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Family Intervention - Proportion of Daily Tasks Completed
Description: The proportion of family-based daily tasks successfully completed will be reported
Time Frame: postoperative day one through postoperative day three
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Family Intervention - Length of Time, Stimulating Activity
Description: Cumulative length of time spent on prescribed stimulating activities
Time Frame: postoperative day one through postoperative day three
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Agreement - FAM-CAM and Research-based CAM Assessments
Description: Agreement will be assessed, via Cohen's kappa, between FAM-CAM and research-based CAM assessments.
Time Frame: postoperative day one through postoperative day three
Reporting Status: Not Posted

19. Other Pre Specified Outcome: 30-Day FAM-CAM Assessments
Description: Incidence (%) of positive FAM-CAM assessments post-discharge
Time Frame: day after discharge through 30 days postoperatively
Reporting Status: Not Posted

20. Other Pre Specified Outcome: 36-Item Short Form Survey
Description: Comprehensive survey that reports on overall health, functional status, physical/mental well-being, and pains (score range, for both overall scale and domain subscales: n, 0-100, 0 = worst score and 100 = best score in relation to the general state of health and quality of life)
Time Frame: 30 days after hospital discharge
Reporting Status: Not Posted

21. Other Pre Specified Outcome: PROMIS Cognitive Abilities (Short Form 4a)
Description: Subjective reporting of cognitive function
Time Frame: 30 days postoperatively
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Hospital Readmission
Description: Incidence (%) of hospital readmission
Time Frame: within 30 days after discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for up to 30 days after surgery.
Arm/Group | Usual Care Group | HELP Support System | Family Support System | Combined Support Systems
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/12 | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 3/15 | 6/12 | 2/14 | 1/16
Other Adverse Events (participants affected / at risk) | 3/15 | 2/12 | 3/14 | 3/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Group (N=15) | HELP Support System (N=12) | Family Support System (N=14) | Combined Support Systems (N=16)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bowel Injury (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C. Difficile (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Difficulty Swallowing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Unresponsive (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Group (N=15) | HELP Support System (N=12) | Family Support System (N=14) | Combined Support Systems (N=16)
Cough, Shortness of Breath, Penile Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental Status Change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Concern for healthcare associated pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left-sided facial droop (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis of left lower leg (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT04007523/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT04007523/ICF_000.pdf